CLINICAL TRIAL: NCT00225615
Title: A Phase 3, Multicenter, Open-Label Extension Study of Phenoptin in Subjects With Phenylketonuria Who Have Elevated Phenylalanine Levels
Brief Title: A Phase 3, Multicenter, Open-Label Extension Study of Phenoptin in Subjects With PKU Who Have Elevated Phenylalanine Levels
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: BioMarin Pharmaceutical (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PKU-004
Record Dates: First submitted 2005-09-22; First posted 2005-09-26 (Estimated); Last update posted 2009-08-20 (Estimated); Status verified 2009-08

CONDITIONS: Phenylketonurias
Keywords: Phenylalanine Hydroxylase
MeSH Terms: conditions — Phenylketonurias | interventions — sapropterin

INTERVENTIONS:
Drug: sapropterin dihydrochloride

SUMMARY:
The primary objective of this trial is to evaluate the safety and tolerability of long-term Phenoptin treatment in subjects with PKU.

ELIGIBILITY:
Inclusion Criteria:

* 8 years of age and older
* Prior successful participation in Study PKU-003
* Willing and able to provide written informed consent or assent and written informed consent (if required) by a parent or legal guardian
* For females of child-bearing potential only: Negative urine pregnancy test within 24 hours prior to enrollment. Women using acceptable birth control measures must agree to continue to use those measures while participating in the study
* Willing and able to comply with study procedures
* Willing to continue current diet unchanged while participating in the study

Exclusion Criteria:

* Perceived to be unreliable or unavailable for study participation or, if under the age of 18, have parents or legal guardians who are perceived to be unreliable or unavailable
* Withdrew from, or otherwise did not successfully complete, study PKU-003, except for subjects who were removed from the study because their blood Phe exceeded the alert level
* Expected to require any investigational agent or vaccine prior to completion of all scheduled study assessments
* Pregnant or breastfeeding, or planning pregnancy
* Concurrent disease or condition that would interfere with study participation or safety (e.g., seizure disorder, oral steroid-dependent asthma or other condition requiring oral or parenteral corticosteroid administration, or insulin-dependent diabetes)
* Requirement for concomitant treatment with any drug known to inhibit folate synthesis (e.g., methotrexate)
* Concurrent use of levodopa

Min Age: 8 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 100
Dates: Start 2005-11; Study Completion 2006-06 (Actual)

PRIMARY OUTCOMES:
Primary objective:
- To evaluate the safety and tolerability of long-term Phenoptin treatment in subjects with PKU.

SECONDARY OUTCOMES:
Secondary objectives:
To compare the safety and tolerability of three different doses of Phenoptin treatment in subjects with PKU.
To determine the effect of various doses of Phenoptin on blood phenylalanine (Phe) levels.
To evaluate the population pharmacokinetics of Phenoptin.
To evaluate the ability of Phenoptin to reduce phenylalanine (Phe) levels over a 24-hour period.
To evaluate the persistence of benefit of Phenoptin treatment in the subject population as evidenced by long-term control of blood Phe levels.

CONTACTS AND LOCATIONS:
Overall Officials: Alex Dorenbaum, MD, Study Chair — BioMarin Pharmaceutical
Locations (14):
- United States (14):
  - Los Angeles, California
  - Oakland, California
  - Sacramento, California
  - San Jose, California
  - New Haven, Connecticut
  - Atlanta, Georgia
  - Chicago, Illinois
  - Minneapolis, Minnesota
  - St Louis, Missouri
  - New York, New York
  - Portland, Oregon
  - Dallas, Texas
  - Salt Lake City, Utah
  - Madison, Wisconsin